CLINICAL TRIAL: NCT05513183
Title: A Phase II Trial to Analyze Clinical and Pharmacological Properties for Severe Neutropenia After Cytoreductive Surgery Followed by Hyperthermic Intraperitoneal Chemotherapy Using Mitomycin-C
Brief Title: Severe Neutropenia After HIPEC Using Mitomycin-C
Status: Completed | Type: Observational
Sponsor: Gangnam Severance Hospital (Other)
Responsible Party: Principal Investigator, Eun Jung Park, Assistant Professor, Gangnam Severance Hospital
Other Study IDs: 3-2021-0122
Record Dates: First submitted 2022-08-18; First posted 2022-08-24 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-08

CONDITIONS: Colorectal Cancer Metastatic; Cancer Metastatic to the Peritoneal Cavity; Appendiceal Neoplasm; Pseudomyxoma Peritonei
MeSH Terms: conditions — Appendiceal Neoplasms; Pseudomyxoma Peritonei

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Peritoneal fluid and plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Arm I (Severe neutropnia group),: After CRS followed by HIPEC using MMC of 35mg/m2, patients who had absolute neutrophil count (ANC) < 1000/mm3 during the postoperative period are assigned as experimental group (Arm I, severe neutropnia group).
  Interventions: Procedure: Intraoperative blood and peritoneal fluid samplings during HIPEC
- Arm II (No severe neutropenia group): After CRS followed by HIPEC using MMC of 35mg/m2, patients who had ANC ≥ 1000/mm3 during the postoperative period are assigned as the control group (Arm II: no severe neutropenia group).
  Interventions: Procedure: Intraoperative blood and peritoneal fluid samplings during HIPEC

INTERVENTIONS:
Procedure: Intraoperative blood and peritoneal fluid samplings during HIPEC — - Intraoperative samplings of blood and peritoneal fluids during HIPEC :
  * Blood sampling of 5ml at each time point (baseline, 0 (HIPEC starting point), 15, 30, 45, 60, 75, 90, 120 min)
  * Peritoneal fluid sampline of 5ml at each time point (baseline, 0 (HIPEC starting point), 15, 30, 45, 60, 75, 90 min)

SUMMARY:
Mitomycin-C (MMC) is the most commonly used chemotherapeutic agent for hyperthermic intraperitoneal chemotherapy (HIPEC) after cytoreductive surgery (CRS) to treat colorectal cancer patients with peritoneal metastases. However, MMC has a side effect of myelosuppression. Particularly, severe neutropenia after CRS with HIPEC can be a life-threatening condition. Despite the postoperative risks of this side effect, the causes and risk factors for severe neutropenia after CRS followed by HIPEC is not identified so far. Therefore, in this study, we aimed to evaluate to evaluate clinical risk factors and pharmacologic properties after CRS with HIPEC using MMC in patients with colorectal cancer or appendiceal mucinous neoplasms with peritoneal metastases.

DETAILED DESCRIPTION:
Evaluation parameters

1. Preoperative period

   * Obtaining informed consent
   * Assessment of baseline clinical characteristics: vital sign, BMI, BSA, ASA classification, ECOG, CBC, CEA level
   * Before 1 day of surgery, assessment of QoR-40 questionnaires
2. Intra-operative period

   * CRS / HIPEC
   * Assessment for peritoneal cancer index, complete cytoreduction score
   * HIPEC procedures: HIPEC was performed using MMC 35 mg/m2 at 41-43℃ for 90 min. Following the HIPEC triple method, MMC 35 mg/m2 was mixed with 3L of Physioneal PD-2 1.5% peritoneal dialysis solution and administered into the intraperitoneal cavity at 50% of the dose at the beginning of HIPEC, 25% of the dose at 30 min, and 25% of the dose at 60 min.
   * Intraoperative samplings of blood and peritoneal fluids during HIPEC :

     * Blood sampling of 5 ml at each time point (baseline, 0 (HIPEC starting point), 15, 30, 45, 60, 75, 90, 120 min)
     * Peritoneal fluid sampling of 5 ml at each time point (baseline, 0 (HIPEC starting point), 15, 30, 45, 60, 75, 90 min)
3. Postoperative period : Postoperative assessment until the discharge date or postoperative 14th days.

   * Daily assessment before discharge : vital sign, transfusion, neutropenia occurrence, adverse events, hematologic blood test (CBC, absolute neutrophil count (ANC), postoperative complications, use of G-CSF, ICU admission (If severe neutropenia occurs in the postoperative period, the patient assigns in arm I.)
   * CEA level: postoperative 5th day
   * QoR-40 questionnaires: postoperative 4th and 7th days

ELIGIBILITY:
Inclusion Criteria:

* Joined the study voluntarily and signed informed consent form
* Patients who diagnosed colorectal cancer or appendiceal mucinous neoplasm with peritoneal metastases
* Patients who undergo CRS/HIPEC using MMC
* ECOG ≤ 1

Exclusion Criteria

* Patients who received synchronous operations for liver or lung metastatic sites during CRS/HIPEC
* Previous histories who underwent CRS/HIPEC
* Patients who received palliative 3rd line chemotherapy
* Patients who received chemotherapy within 1 year to treat other cancers
* Patients who had PCD cathethers for ascites control
* ECOG ≥2
* Infectious status
* Age<19 years old
* Pregnant or breast-feeding women or people during the birth-period who refused to take contraceptives

Drop-out criteria

- Hospital stay > 30 days

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who diagnosed colorectal or appendiceal neoplasms with peritoneal metastases who underwent cytoreductive surgery and hyperthermic intraperitoneal chemotherapy using mitomycin-C
Sampling Method: Non-Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2021-05-20 (Actual); Primary Completion 2023-03-20 (Actual); Study Completion 2023-03-20 (Actual)

PRIMARY OUTCOMES:
Association between the concentration of intraoperative mitomycin-C absoprtion and severe neutropenia after CRS/HIPEC | 2 weeks after the discharge
  Comparison of the pharmacologic association between occurrence of postoperative severe neutropenia, and blood absoprtion rates of MMC and the area-under-the curve (AUC) ratios during HIPEC

SECONDARY OUTCOMES:
Incidence of severe neutropenia | During 2 weeks after CRS/HIPEC
  Incidence (rates)
Postoperative complications | During 2 weeks after CRS/HIPEC
  Assessment from Clavien-Dindo classification
Patterns of perioperative changes of WBC, Hemoglobin, platelet, lymphocyte, neutrophil counts | During 2 weeks after CRS/HIPEC
  Records for serologic tests
Frequency of postoperative uses for G-CSF | During 2 weeks after CRS/HIPEC
  Numbers of G-CSF uses
Changes of CEA level | During 2 weeks after CRS/HIPEC
  ng/mL
Quality of Life: QoR-40 questionnaire | During 2 weeks after CRS/HIPEC
  Answer of questionnarie

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Colon and Rectal Surgery, Department of Surgery, Gangnam Severance Hospital, Yonsei University College of Medicine, Seoul, South Korea, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Verwaal VJ, van Ruth S, de Bree E, van Sloothen GW, van Tinteren H, Boot H, Zoetmulder FA. Randomized trial of cytoreduction and hyperthermic intraperitoneal chemotherapy versus systemic chemotherapy and palliative surgery in patients with peritoneal carcinomatosis of colorectal cancer. J Clin Oncol. 2003 Oct 15;21(20):3737-43. doi: 10.1200/JCO.2003.04.187. PMID 14551293
- [Background] Katz MH, Barone RM. The rationale of perioperative intraperitoneal chemotherapy in the treatment of peritoneal surface malignancies. Surg Oncol Clin N Am. 2003 Jul;12(3):673-88. doi: 10.1016/s1055-3207(03)00034-6. PMID 14567024
- [Background] Kuzuya T, Yamauchi M, Ito A, Hasegawa M, Hasegawa T, Nabeshima T. Pharmacokinetic characteristics of 5-fluorouracil and mitomycin C in intraperitoneal chemotherapy. J Pharm Pharmacol. 1994 Aug;46(8):685-9. doi: 10.1111/j.2042-7158.1994.tb03883.x. PMID 7815285
- [Background] Lambert LA, Armstrong TS, Lee JJ, Liu S, Katz MH, Eng C, Wolff RA, Tortorice ML, Tansey P, Gonzalez-Moreno S, Lambert DH, Mansfield PF. Incidence, risk factors, and impact of severe neutropenia after hyperthermic intraperitoneal mitomycin C. Ann Surg Oncol. 2009 Aug;16(8):2181-7. doi: 10.1245/s10434-009-0523-4. Epub 2009 May 28. PMID 19475451
- [Background] Feferman Y, Bhagwandin S, Kim J, Aycart SN, Feingold D, Labow DM, Sarpel U. Conflicting Data on the Incidence of Leukopenia and Neutropenia After Heated Intraperitoneal Chemotherapy with Mitomycin C. Ann Surg Oncol. 2017 Dec;24(13):3831-3836. doi: 10.1245/s10434-017-6112-z. Epub 2017 Oct 12. PMID 29027153
- [Background] Park EJ, Lee SJ, Baik SH. ASO Author Reflections: Delayed Occurrence and Postoperative Risks of Mitomycin-C-Induced Neutropenia After Hyperthermic Intraperitoneal Chemotherapy. Ann Surg Oncol. 2022 Mar;29(3):2087-2088. doi: 10.1245/s10434-021-11000-2. Epub 2021 Oct 23. No abstract available. PMID 34689262
- [Background] Lee SJ, Jeon Y, Lee HW, Kang J, Baik SH, Park EJ. Impact of Mitomycin-C-Induced Neutropenia after Hyperthermic Intraperitoneal Chemotherapy with Cytoreductive Surgery in Colorectal Cancer Patients with Peritoneal Carcinomatosis. Ann Surg Oncol. 2022 Mar;29(3):2077-2086. doi: 10.1245/s10434-021-10924-z. Epub 2021 Oct 19. PMID 34665362